CLINICAL TRIAL: NCT02242994
Title: Data Acquisition Study for a Communication Device for Pediatric Patients With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Axel Krieger (Other)
Responsible Party: Sponsor-Investigator, Axel Krieger, MD, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00003767
Record Dates: First submitted 2014-07-24; First posted 2014-09-17 (Estimated); Results first posted 2016-12-14 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-10

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

ARMS (1):
- Dynavox Maestro and Experimental App (Experimental): Receives both Experimental App and Dynavox Maestro to communicate. Each participant will receive both devices. Order of device received is randomly assigned.
  Interventions: Device: Dynavox Maestro; Device: Experimental App

INTERVENTIONS:
Device: Dynavox Maestro — Receives commercially available communication device Dynavox Maestro to test speed and quality of communication.
Device: Experimental App — Participant receives experimental app to test speed and error rate of communication.

SUMMARY:
The purpose of this study is to evaluate a touch screen application designed to help pediatric patients with cerebral palsy communicate. The study will test how well patients type on two different tools: one tool is already on the market , and the second tool is a newly developed App.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 7 years old - 21 years old
* been diagnosed with spastic or dystonic diplegic or quadriplegic cerebral palsy.
* are able to communicate through written words
* are able to follow a 3- steps directions, and follow study directions and procedures.

Exclusion Criteria:

-

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2014-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's National, Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dynavox Maestro and Experimental App
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Age 7-21
Arm/Group | Dynavox Maestro and Experimental App
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.6 (4.3)
Gender [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Speed of Communication
Description: Measure time (in minutes) to type 3 pre-set sentences
Time Frame: Immediately
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Dynavox Maestro and Experimental App
Number analyzed (Participants) | 5
minutes
  Experimental App | 8.13 (12.61)
  Dynavox | 2.96 (4.28)

2. Secondary Outcome: Error Rate of Communication
Description: Amount of typing errors per sentence
Time Frame: At time of experiment
Measure: Mean (Standard Deviation); unit: errors
Arm/Group | Dynavox Maestro and Experimental App
Number analyzed (Participants) | 5
errors
  Experimental App | 0.12 (0.45)
  Dynavox | 0.11 (0.40)

ADVERSE EVENTS:
Arm/Group | Dynavox Maestro and Experimental App
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes